CLINICAL TRIAL: NCT01570647
Title: Automated Connective Tissue Torque Sensor
Acronym: StromaTorque
Status: Completed | Type: Observational
Sponsor: Stromatec, Inc. (Industry)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Robert Davis, Principal Investigator, Stromatec, Inc.
Other Study IDs: R44AT004379 (NIH)
Record Dates: First submitted 2012-04-01; First posted 2012-04-04 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Connective Tissue; Musculoskeletal Pain
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- Healthy controls
- Chronic low back pain
- restricted hamstrings
- systemic scleroderma
- joint hyperlaxity

SUMMARY:
The purpose of this study is to develop a measure - the needle torque test - capable of detecting connective tissue abnormalities associated with musculoskeletal disorders.

DETAILED DESCRIPTION:
Chronic musculoskeletal pain is a source of considerable disability, work absenteeism and health care costs. A major obstacle to the treatment of these conditions is the lack of methods to objectively assess connective tissues and measure the effect of treatments. Needle torque test technology under development in this project will potentially enable objective measurement of connective tissue abnormalities associated with musculoskeletal pain and dysfunction. This could help evaluate the efficacy of various treatments and enhance the objective monitoring of patient progress in clinical practice.

ELIGIBILITY:
Inclusion Criteria for chronic low back pain subjects:

* back pain that has disrupted activity for more than half the days in the past 12 months.

Inclusion Criteria for restricted hamstring subjects:

* 90/90 test of more than 20 degrees

Inclusion Criteria for systemic scleroderma subjects:

* physician diagnosis

Inclusion criteria for joint hyperlaxity subjects:

* Beighton test score of 7 or higher

Exclusion Criteria for all subjects:

* surgery or scars in thighs or low back
* neurological or major psychiatric disorder
* bleeding disorders
* acute systemic infection
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2012-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Number of needle revolutions to achieve threshold torque | Time zero, 30 minutes and one week

CONTACTS AND LOCATIONS:
Overall Officials: Robert Davis, Principal Investigator — Stromatec, Inc.
Locations (1):
- Stromatec, Inc., Burlington, Vermont, United States